CLINICAL TRIAL: NCT06124820
Title: A Single-blinded, Randomised Controlled Trial Comparing the Use of Intravaginal Laser Therapy to Sham in Post-menopausal Women with Recurrent Urinary Tract Infections (rUTI) and the Impact on the Vaginal and Urinary Microbiome
Brief Title: RCT Comparing Intravaginal Laser Therapy to Sham in Post-menopausal Women with Recurrent Urinary Tract Infections
Acronym: UTIEXTERMINATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 302037
Record Dates: First submitted 2022-09-06; First posted 2023-11-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Urinary Tract Infection; Genitourinary Syndrome of Menopause
Keywords: UTI; Recurrent Urinary Tract Infection; Genitourinary Syndrome of Menopause; Laser; CO2 Laser; Microbiome
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Monalisa Touch (SmartXide2 V2LR, DEKA, Florence, Italy)
Who Masked: Participant
Masking Description: Sham
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Intravaginal micro-ablative fractional CO2 laser technology Deka SmartXide Touch C60 (MonaLisa Touch) will be administered intravaginally over a course of 5 cycles
  Interventions: Device: Deka SmartXide Touch C60 (MonaLisa Touch)
- Control Arm (Sham Comparator): Sham treatment -Participants receiving sham treatment will have the probes advanced in the same manner without the use of a laser energy device.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Deka SmartXide Touch C60 (MonaLisa Touch) — Intravaginal micro-ablative fractional CO2 laser technology Deka SmartXide Touch C60 (MonaLisa Touch)
  Arms: Treatment Arm
Device: Sham — Participants receiving sham treatment will have the probes advanced in the same manner without the use of a laser energy device.
  Arms: Control Arm

SUMMARY:
Recurrent urinary tract infection (rUTI) is a common and difficult to treat problem with limited treatment option; postmenopausal women are disproportionately affected. The genitourinary syndrome of menopause (GSM) describes the broad spectrum of signs and symptoms caused by the loss of endogenous sex steroids. The combined effects of urogenital epithelial tissue thinning and changes to the vaginal and bladder microbiome can predispose to ascending UTIs. Recurrent UTIs is a component of GSM.

Intravaginal laser therapy has been shown to be safe and effective for the treatment of GSM, however, the role of laser for treatment of recurrent UTIs is unknown. We hypothesis that the incidence of UTI will be reduced as CO2 laser restores vaginal epithelium to a state similar to that of a pre-menopausal woman, preventing microtrauma, and increases Lactobacillus and normal flora (Athanasiou et al., 2016). Lactobacillus is considered the bacteria that helps keep the vagina healthy and infection free through its production of lactic acid which lowers vaginal pH, this more acidic environment may be protective from uropathogens.

We therefore aim to conduct a single-blinded, multi-centre, randomised controlled trial comparing the use of intravaginal CO2 laser therapy to sham in post-menopausal women with rUTIs and to determine the impact on the microbiome.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are the most common outpatient infection with a prevalence of 20% in women over 65, compared with 11% in the overall population (Chu and Lowder, 2018).

The genitourinary syndrome of menopause (GSM) is the accepted term used to describe the broad spectrum of genitourinary tract symptoms and signs caused by the loss of endogenous sex steroids that occurs at the time of and after the menopause. Global improvements in healthcare have resulted in an aging population. Today women are spending 40% of their lives in the postmenopausal state with 50-70% of postmenopausal women reporting symptomatic GSM. The combined effects of urogenital epithelial tissue thinning and changes to the vaginal and bladder microbiome can predispose to ascending UTIs. Recurrent UTIs is a component of GSM.

Current interventions for recurrent urinary tract infections in women include lifestyle and behavioural advice, complimentary therapies and antibiotics. These treatment regimens are not always effective or acceptable. Intravaginal Laser therapy is an alternative non-hormonal treatment of GSM as it stimulates tissue repair and restores normal vaginal function.

Currently intravaginal laser therapy has been shown to be safe and effective for the treatment of GSM, as described in a recent network analysis of 29 randomised controlled studies, incorporating 8311 patients (Li et al., 2021). Provisional results using FemTouch®, fractional CO2 laser, appear promising with 9/12 (75%) of post-menopausal women UTI free at 12 months follow-up (Yang and Foley). However, there is a scarcity of studies available looking at the impact of this novel technology for the treatment of recurrent UTIs.

The investigators aim to conduct a single-blinded, randomised controlled trial comparing the use of intravaginal CO2 laser therapy to sham in post-menopausal women with rUTIs and to determine the impact on the microbiome. The investigators hypothesise that this treatment will be effective in reducing the incidence of urinary tract infection as CO2 laser through a process of thermomodulation, simulates tissue repair by restoring vaginal epithelium to a state similar to that of a pre-menopausal woman. In addition, a study assessing the effect of micro-ablative functional CO2 laser reported an increase in Lactobacillus and normal flora (Athanasiou et al., 2016). Lactobacillus is considered the bacteria that helps keep the vagina healthy and infection free through its production of lactic acid which lowers the vaginal pH, this more acidic environment may be protective from uropathogens. The role and impact of Laser on other microbial communities is still not fully understood, this study aims to expand this knowledge base.

Recurrent UTIs is a common and difficult to treat problem with limited treatment options, this study endeavors to expand the knowledge pool and provide alternative non-pharmacological options using this novel technology.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* History of recurrent UTI (Defined as women who have suffered at least three episodes of symptomatic UTI within the preceding 12 months or two episodes in the last six months, or at least one episode of UTI requiring hospitalisation, or if previously prescribed prophylactic antibiotics for UTI, have completed a 3-month washout period without antibiotic prophylaxis)
* Able to give informed consent for participation in the trial
* Able and willing to adhere to a 17-month study period

Exclusion Criteria:

* Not willing to abstain from vaginal intercourse for 48 hours following laser-therapy
* Use of vaginal hormonal therapy in the three months before study start
* History of a genital fistula, a thin recto-vaginal septum as determined by the investigator or history of a fourth-degree laceration during physical screening exam (e.g., deficient perineal body)
* Active sexually transmitted disease upon vaginal exam (as determined by the investigator) that precludes treatment or any other vaginal infection
* History of lichen sclerosis
* History of radiotherapy for cervical or uterine cancer
* A medical condition that may interfere with participants' compliance with the protocol
* Women with correctable urinary tract abnormalities that are considered to be contributory to the occurrence of rUTI
* Women taking Methenamine Hippurate and unable to undergo a three-month washout period
* Undiagnosed genital bleeding
* Women who self-catheterise, or have an indwelling/suprapubic catheter
* Unable to give informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-10-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
To determine and compare the incidence of symptomatic antibiotic-treated UTI during the 6-month follow-up period after completion of allocated treatment | 6 months
  Determined from the UTI history diary and cross-referenced with hospital and GP records

SECONDARY OUTCOMES:
UTI history diary | 18 months
  Participants will be given a UTI history diary to complete which will documents all symptomatic and treated UTI, the diary will be cross-referenced with participant history and review of medical history at each follow-up appointment.
Vaginal Health Index Score (VHIS) | 18 months
  o It incorporates a clinical examination of the vagina for pH, elasticity, fluid volume, epithelial integrity, moisture. Vaginal pH will be obtained using a piece of litmus paper placed on the lateral wall of the vagina.
King's Health Questionnaire (KHQ) | 18 months
  21 items about urinary tract symptoms yield scores in 9 domains (general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy & severity of symptoms).
International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) | 18 months
  A 12 item questionnaire for evaluating female lower urinary tract symptoms
International Consultation on Incontinence Questionnaire - Vaginal Symptoms (ICIQ-VS) | 18 months
  A 14 item questionnaire for evaluating vaginal symptoms, associated sexual matters and impact on quality of life (QoL)
10 cm Visual Analogue Scale for Symptoms (VAS) | 18 months
  Consists of a 10cm line, used to determine intensity of symptoms with two endpoints representing 0 ("no symptoms" and 10 ("symptom at the worse it could be"). Symptoms assessed: vaginal dryness, dyspareunia, itching, burning, dysuria, frequency, urgency, overall symptoms
Urinary Tract Infection Symptom Assessment Questionnaire (UTISA) | 18 months
  14-item questionnaire asking about the severity and bothersome of seven key UTI symptoms.
Female Sexual Function Index Scoring (FSFI) | 18 months
  A 19 item questionnaire designed to measure sexual functioning in women.
Health Service Utilisation Questionnaire (HSU-Q) | 18 months
  An instrument for the standardized and systematic assessment of various aspects of health care utilisation
Treatment satisfaction questionnaire for laser (TSQ-L) | 18 months
  A modified 10-item questionnaire used to determine participant satisfaction with treatment
Vulvoscopic Genital Tissue Appearance Scale (VGTA) | 18 months
  assesses 10 parameters of the appearance of the genital tissue including loss of labia minora/majora, decreased glans clitoris, stenosis of introitus, prominence of the urethral meatus, vestibular pallor, vestibular pallor, vesicular erythema, loss of vaginal rugae, loss of vestibular moisture and loss of prominence of the anterior vaginal wall. A score of 0 to 30 is obtained, the higher the score the worse the vulvoscopic genital tissue appearance
Adverse event recording | 18 months
  Adverse events will be asked at each visit and participant will have contact details to reports any throughout the study period
Dipstick urine analysis | 18 months
  Reagent strips used to detect substances in urine including nitrate, leucocytes, glucose, protein, pH, ketones and blood
Standard urine culture | 18 months
  Routine urinalysis that identify bacteria or yeast causing a urinary tract infection
Expanded Quantitative Urine Culture (EQUC) | 18 months
  - EQUC uses larger urine volume, longer incubation times, multiple growth media and atmospheric conditions and enables species-level identification
16S rRNA rapid Next-generation Gene Sequencing | 18 months
  16S rRNA NGS provide gene-level information for species. It utilises PCR amplification and NGS of essential 16S ribosomal RNA genes. It enables the evaluation of even closely related bacterial species through evolutionary polymorphisms
Shotgun metagenomic sequencing | 18 months
  allows the identification and profiling of microbial species independent of reference sequences.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Will be available at request